CLINICAL TRIAL: NCT02878070
Title: My Care My Call: Peer-Led Health Empowerment Training For People With Chronic Spinal Cord Injury
Brief Title: My Care My Call: Peer-Led Health Empowerment Training in Chronic Spinal Cord Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University (Other)
Collaborators: Gaylord Hospital (Unknown); Hospital for Special Care (Unknown); National Institute on Disability, Independent Living, and Rehabilitation Research (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 90SI5013
Record Dates: First submitted 2016-08-22; First posted 2016-08-25 (Estimated); Last update posted 2016-08-25 (Estimated); Status verified 2016-08

CONDITIONS: Spinal Cord Injuries
Keywords: Spinal Cord Injuries; Telemedicine; Health Behaviors
MeSH Terms: conditions — Spinal Cord Injuries; Health Behavior

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Peer Health Coaching (Experimental): Calls from a Peer Health Coach for 6 months
  Interventions: Behavioral: Calls from a Peer Health Coach for 6 months
- Usual Care (No Intervention)

INTERVENTIONS:
Behavioral: Calls from a Peer Health Coach for 6 months — Weekly calls for 2 months, bi-weekly calls for 2 months, monthly calls for 2 months.
  Arms: Peer Health Coaching

SUMMARY:
My Care My Call (MCMC) is an innovative, peer-led telephone intervention designed to empower adults with chronic spinal cord injury (SCI) in the self-management of their primary health care needs to prevent secondary conditions. In a randomized controlled trial, participants assigned to the MCMC intervention receive tapered calls from a Peer Health Coach (PHC) for six months. PHCs are experienced, empathetic peer mentors living with SCI who act as supporters, role models, and advisors, providing goal-setting support, motivation, education, and resource referral to participants. Participants complete surveys at baseline, 2, 4, and 6-months, as well as qualitative exit phone interviews.

It is hypothesized that MCMC will: 1) Increase participants' self-advocacy in health care interactions as reflected in increases in three domains of self-advocacy: assertiveness, illness education, and potential for mindful non-adherence, 2) Increase participants' self-efficacy for health care navigation, preference for involvement in, and satisfaction with their primary care physician (PCP), and 3) Increase health related quality of life and medical social support compared with those receiving usual care. Additional secondary hypotheses state that the MCMC intervention will increase access to primary care and use of preventive screening services compared with those receiving usual care.

ELIGIBILITY:
Inclusion Criteria:

* Self-report of physician-confirmed traumatic spinal cord injury diagnosis
* Injured one year ago or more
* Telephone access for at least 9 months
* Speaks and understands conversational English
* Have a current health issue to address

Exclusion Criteria:

* Moderate to severe cognitive impairment
* Surgery scheduled for a 2-week or longer duration during the months of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2015-01; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Patient Activation Measure (PAM) | Change in PAM score from baseline to 2, 4, and 6 months
  Measurement of self-management behavior

SECONDARY OUTCOMES:
Patient Self-Advocacy Scale (PSAS) | Change in PSAS score from baseline to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Alan Jette, PT, PhD, Principal Investigator — Boston University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Houlihan BV, Brody M, Everhart-Skeels S, Pernigotti D, Burnett S, Zazula J, Green C, Hasiotis S, Belliveau T, Seetharama S, Rosenblum D, Jette A. Randomized Trial of a Peer-Led, Telephone-Based Empowerment Intervention for Persons With Chronic Spinal Cord Injury Improves Health Self-Management. Arch Phys Med Rehabil. 2017 Jun;98(6):1067-1076.e1. doi: 10.1016/j.apmr.2017.02.005. Epub 2017 Mar 8. PMID 28284835